CLINICAL TRIAL: NCT00365573
Title: Doppler Ultrasonography Evaluation of Tibial Fracture Site Vascularity
Status: Suspended | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: USTF001-HMO-CTIL
Record Dates: First submitted 2006-08-16; First posted 2006-08-17 (Estimated); Last update posted 2010-11-05 (Estimated); Status verified 2010-10

CONDITIONS: Tibial Fracture
MeSH Terms: conditions — Tibial Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to evaluate the blood supply to patients that are suffering from fracture in the tibia by UltraSound Doppler.

ELIGIBILITY:
Inclusion Criteria:

* Above 16 years old

Exclusion Criteria:

* Pregnancy

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patient witj tibial fracture.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-02

CONTACTS AND LOCATIONS:
Overall Officials: Ori Safran, Dr., Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel